CLINICAL TRIAL: NCT06310655
Title: A Novel Pilot Study of Online Proton Adaptive RadioTherapY (PARTy) Utilizing Computed Tomography On Rails
Brief Title: Online Proton Adaptive Radiotherapy
Acronym: PARTy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202403078
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor
Keywords: SBRT; proton radiotherapy; reirradiation; Adaptive radiation therapy; Online adaptive radiotherapy; online proton adaptive radiotherapy

STUDY DESIGN:
Intervention Model Description: All patients will receive 5 fractions of proton radiotherapy for their cancer. At the time of each fraction, the initial pre-plan will be compared to the newly generated adapted plan, and the optimal treatment will be administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Proton Stereotactic Body Radiotherapy (SBRT) (Experimental): All patients will receive standard of care proton SBRT either daily or every other day for a total of 5 fractions. At the time of each treatment, the initial pre-plan will be generated on the patient and assessed for coverage and safety. An adaptive plan based on the patient's anatomy that day will also be generated and then compared to the initial pre-plan. The optimal treatment plan will be chosen and administered to the patient on that day. This process will be repeated for each fraction for every patient.
  Interventions: Radiation: Proton SBRT

INTERVENTIONS:
Radiation: Proton SBRT — Patients will receive SBRT over 5 days, either every day or every other day, to a dose of 25-50 Gy.

SUMMARY:
This is a pilot study evaluating the feasibility of daily online adaptive planning for patients undergoing proton radiation therapy.

Patients undergoing proton radiation therapy normally undergo extensive pre-planning for their treatment. However, accounting for uncertainties in treatment delivery remains a challenge for a variety of reasons, such as differences in patient anatomy from pre-planning to the day of treatment. Online adaptive planning is a process consisting of generating the original pre-plan on the patient on a treatment day, assessing the pre-plan's coverage and safety, and if changes are needed, the plan is changed in order to optimize the treatment while the patient is still on the treatment table. This study is assessing the feasibility and safety of this approach in order to gather data for a larger trial.

ELIGIBILITY:
Inclusion Criteria:

* Oligometastatic or primary malignancy planned for proton SBRT. Disease site should be biopsy-proven primary disease of solid tumor histology with the exception of Hepatocellular carcinoma (HCC). HCC does not need to be biopsy proven if imaging and clinical findings are consistent with the diagnosis.
* Must be deemed medically fit for proton SBRT by the treating physician.
* Prior radiation therapy is allowed.
* At least 18 years of age.
* Karnofsky ≥ 70%.
* Because radiation therapy is known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, or a male suspect he has fathered a child, s/he must inform the treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Histology of small cell carcinoma. Mixed histologies with a predominantly small cell component are also exclusionary.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Medical contraindication to proton therapy or any other condition that in the opinion of the treating radiation oncologist, renders the patient unfit for SBRT
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum or urine pregnancy test within 14 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Feasibility of online proton adaptive radiotherapy | Through end of treatment (up to 2 weeks)
  Feasibility will be defined as successful completion of the online adaptive proton radiotherapy workflow in at least 70% of planned adaptive fractions.

SECONDARY OUTCOMES:
Safety of online proton adaptive radiotherapy as measured by the amount of grade 2 and higher radiation-related toxicities | from start of treatment through 3 months
  Adverse events are graded per CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Waters, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this trial after de-identification. Other documents may be shared include the study protocol.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months after article publication.
Access Criteria: Proposals to access study data should send request to amo@wustl.edu. To gain access, data requesters must sign data access agreement.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu